CLINICAL TRIAL: NCT04984083
Title: Maternal and Neonatal Benefits of Prophylactic Administration of Vitamin K Before Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Faculty of Medicine, Minia University (Unknown)
Responsible Party: Principal Investigator, Mazen Abdel Rasheed, Researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Prophylactic Vitamin K
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Vitamin K
MeSH Terms: interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): patients will take vitamin k 10 mg/ml once daily orally or IM between four and 96 hours before elective cesarean section
  Interventions: Dietary Supplement: vitamin k
- Group II (No Intervention): patients will not take vitamin k before cesarean section

INTERVENTIONS:
Dietary Supplement: vitamin k — patients will take vitamin k 10 mg/ml once daily orally or IM between four and 96 hours before elective cesarean section
  Arms: Group I

SUMMARY:
Vitamin K deficiency can cause serious risks to pregnant women and their babies that may lead to hemorrhage, especially in newborns. We aim to evaluate the efficacy of vitamin k in decreasing blood loss during and after elective cesarean section (CS), and to assess the neonatal beneficial effects of prophylactic maternal vitamin k administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20-40 years.
2. Gestational age between 36-39 weeks.
3. Patients who will undergo an elective cesarean section.
4. Full-term alive baby.
5. Non-scarred uterus.
6. No obstetric or medical complications.
7. No bleeding tendency.

Exclusion Criteria:

1. Patients at less than 36 gestational weeks.
2. Patient refusal.
3. Patients who have thrombo-embolic complications.
4. Patients with obstetric and medical complications.
5. Patients with anomalous fetuses.
6. Patients on anti-coagulant drugs, long-term antibiotics, and anti-epileptic drugs.
7. Patients with obstetric cholestasis.
8. Patients with a previous history of preterm labor.
9. Patients with multiple pregnancies.
10. Gestational hypertension or preeclampsia.
11. Blood clotting disorders.
12. Placental abnormalities such as, Placenta accreta, Placenta increta, and Placenta percreta.
13. Placental abruption and Placenta previa.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Blood loss (measured in cc) | During Cesarean Section
Prothrombin time of the mother (measured in seconds) | 6 hour postmartum
Activated Partial Thromboplastin Time (APTT) of the mother (measured in seconds) | 6 hour postmartum
Prothrombin Concentration (PC) of the mother (measured in %) | 6 hour postmartum
Prothrombin time of the newborn (measured in seconds) | immediately after birth
Prothrombin Concentration (PC) of the newborn (measured in %) | immediately after birth

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Egypt